CLINICAL TRIAL: NCT04222556
Title: Evaluation of an Optimized Intervention to Prevent Early Substance Use Among American Indian Youth: Examination of Expanded Impacts on Youth and Parents
Brief Title: Evaluation of Thiwáhe Gluwáš'Akapi Substance Use Prevention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 18-2559; R37DA047926 (NIH)
Record Dates: First submitted 2019-11-27; First posted 2020-01-10 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Substance Use; Substance Abuse; Suicide
Keywords: American Indian; Adolescent; Parenting; Family; Prevention
MeSH Terms: conditions — Substance-Related Disorders; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiwáhe Gluwáš'akapi (Experimental): Weeks 1-7: Weekly in-person 2.5 hour family sessions 30 minute family meal 1 hour separate youth and adult sessions
  1 hour family session
  Interventions: Behavioral: Thiwáhe Gluwáš'akapi
- Woyute Waśte (Active Comparator): Respect for community and cultural values regarding research protocols precluded use of a randomized controlled design with a control group receiving no intervention, so we identified a cost-effective comparison condition program to offer value to study participants. A focus on healthy eating and exercise was of interest to community partners and not expected to directly confound the primary outcomes of the TG program (substance use and suicide risk).
  Week 1 in-person 2.5 hour family session 30 minute family meal 2 hour interactive family session (3 stations) Weeks 2-7: text messages with program content and questions
  Interventions: Behavioral: Woyute Waśte

INTERVENTIONS:
Behavioral: Thiwáhe Gluwáš'akapi — Thiwáhe Gluwáš'akapi (TG, sacred home in which family is made strong) is a cultural adaptation of the Strengthening Families Program for Parents and Youth 10-14 (SFP 10-14). TG, like SFP 10-14, is a 7-week family-based prevention program with separate youth and adult sessions followed by family sessions. Videos teach content and spark discussion; games and activities foster interaction and provide opportunities to practice skills. Four key adaptations were made to create TG: (1) cultural kinship teachings and tribal language kinship words were embedded throughout; (2) a parent session on coping with stress was enhanced to teach recognizing and responding to trauma reactions in youth; (3) a session on listening was moved earlier in the curriculum, given cultural oral tradition; (4) session videos were remade with local actors and adapted scenarios. A multiphase optimization strategy design was used to test potential adaptations, resulting in the optimized TG program.
  Arms: Thiwáhe Gluwáš'akapi
Behavioral: Woyute Waśte — Woyute Waśte (WW) was adapted from the Colorado School of Public Health's Integrated Nutrition Education Program (INEP) for the culture and context of the reservation. Families will meet for 1 session to participate in hands-on activities - preparing healthy meals, family physical activity, and sugary drinks. They will discuss setting healthy goals and tracking progress, receive recipes and water bottles, and for 6 weeks after the session, will get text messages with additional program content.
  Arms: Woyute Waśte

SUMMARY:
Researchers at the Centers for American Indian and Alaska Native Health in the Colorado School of Public Health at the University of Colorado completed an intensive community-engaged process to rigorously adapt the Strengthening Families Program for Parents and Youth 10-14 for the cultural context of a Northern Plains reservation community, creating a program optimized for American Indian families, Thiwáhe Gluwáš'akapi (TG, sacred home in which family is made strong). This study will test the effectiveness of TG for delaying the onset of substance use among young adolescents. In response to requests from participating families and community partners to help address suicide risk among their youth, and based on preliminary evidence that the program may impact risk behaviors beyond substance use, the study will also test suicide risk outcomes among youth. Finally, in recognition of the potential for reciprocal influence on the adults participating in the program with their children, capitalizing on their motivation to make concomitant positive changes in their own lives, the current study will also examine effects on adult substance use. In summary, this study will test the effectiveness of TG for reducing risk for: (1) substance use among youth; (2) suicide risk among youth; and (3) substance abuse among adults.

DETAILED DESCRIPTION:
Study design overview

All 13 middle schools on the reservation will participate in this study by providing space for program groups to meet in the evenings and allowing recruitment activities at school events. A total of 480 families will be recruited into 6 cohorts across two years (spring, summer and fall). In each community, families with a child 10-12 years of age will be recruited to participate in the study. Half of recruited families will be randomly assigned to receive the Thiwáhe Gluwáš'akapi (TG) substance use prevention program and half to the comparison group, which will receive the Woyute Waśte (WW) healthy eating and exercise program. Randomization will be explained to families as part of the recruitment and consent process. Given the potential for contamination across groups with this design, the investigators will carefully examine outcomes across groups and statistically control for contamination effects as necessary. Alternative designs, including randomization at the school/community level, were rejected due to greater concerns about cross-community variability.

Recruitment and retention strategies

Schools (e.g., registration, family nights, parent-teacher conferences, holiday events) will be the main points of recruitment but additional advertising and promotion will take place at community events such as powwows, health fairs, and basketball tournaments. Written materials about the program will be distributed, along with promotional items (e.g., water bottles, magnets, and lanyards with the project name and logo). The investigators will also advertise on local community radio, which has wide reach on the reservation. Because TG has been implemented at 12 of the 13 middle schools on the reservation as a part of the adaptation study and has been well received by both families and school staff, the investigators often have inquiries about opportunities for future participation, and anticipate a positive response to recruitment efforts.

Facilitators will call families weekly to touch base with them and remind them about upcoming sessions. The investigators provide meals to families at the start of each program session, giving them opportunities to connect with other families and facilitators, fostering relationships, and making it easier for busy families to get to the sessions. Child care and transportation will be provided, as needed.

Approaches to ensuring fidelity

All facilitators will be trained in TG by a master SFP 10-14 trainer from Iowa State University (Beth Fleming) and the master TG trainer (Dr. Alicia Mousseau, who led the program adaptation). Weekly supervision and preparation for sessions before and during implementation will be provided onsite by local staff certified as TG trainers, who will also train new facilitators as needed due to staff turnover. These on-site trainers will also conduct regular fidelity checks (observations during sessions using standardized fidelity checklists) and provide feedback to facilitators.

Data collection schedule and estimated sample sizes across waves

In each family, up to 2 eligible youth (aged 10-12) and 1 parent/caregiver will be eligible to participate in the research and take study surveys. Sample size estimates for each wave are estimates of the number of families (F), youth (Y), adults (A), and total sample (T). Ranges for youth and total reflect that 1-2 youth per family are eligible to complete surveys. Estimates include an attrition rate of 2.5% every 6 months, based on past experience with families in this community.

1. Baseline - 1-2 weeks before first session: F=480; Y=480-960; A=480; T=960-1440
2. Post-intervention -1 week after last session: F=480; Y=480-960; A=480; T=960-1440 6 follow-up surveys:
3. 6-month: F=468; Y=468-936; A=468; T=936-1404
4. 12-month: F=456; Y=456-912; A=456; T=912-1368
5. 18-month: F=445; Y=445-890; A=445; T=890-1335
6. 24-month: F=434; Y=434-868; A=434; T=868-1302
7. 30-month (excluding final cohort): F=370; Y=370-740; A=370; T=740-1110
8. 36-month (excluding final 2 cohorts): F=206; Y=206-412; A=206; T=412-618

Data collection procedures

All surveys will be administered online, using REDCap survey software. The baseline survey will be collected during an in-person meeting, after consent is obtained, using iPads provided by research staff. Post-intervention surveys will also be administered in person. For follow-up surveys, participants will be sent unique links to access their surveys on their own devices (e.g., computers, phones, tablets) or at a location of their choice (e.g., tribal college center). They will also be able to request to have research staff meet with them to collect these follow-up surveys in person and provide a project iPad for survey completion. Surveys collected via REDCap will be immediately uploaded to a secure cloud storage. REDCap is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. REDCap is hosted by the University of Colorado Anschutz Medical Campus and supported by the Colorado Clinical and Translational Sciences Institute.

Analytic Plan

Three analytic approaches will be used: (1) discrete-time time survival analysis (DTSA), (2) mixed model analyses (MM), and (3) latent growth curve modeling (LGCM). Intention to treat principles will be applied in all analyses. Participant sex will be included as a covariate or separate models will be estimated by gender to explore differential effect patterns. Sandwich-estimators (type=complex in Mplus) and random effects models (in SAS Proc Mixed) will adjust for clustering at the family (and/or school) level. Full information maximum likelihood (FIML) procedures will be used to provide unbiased and efficient estimates.

Discrete-time survival analyses (DTSA) will be used to estimate the probability (hazard) for initiation of substance use among youth who have not used substances prior to enrollment in the study. Initial DTSA analyses will compare the fit of models assuming proportional odds (i.e., constant intervention effect across waves) either with or without frailty (residual variance) to non-proportional odds (i.e., variable intervention effect across waves). Comparisons will be based on the Akaike Information Criterion (AIC) and the Bayesian Information Criterion (BIC). Exposure to TG will be included as a time-invariant covariate to estimate treatment effects on risk of initiation. Mplus Monte Carlo analyses were used to determine power requirements for DTSA models. Effect-size estimates from earlier etiological work in this reservation community were used (hazard age 10-13, alcohol =.14; marijuana = .13, tobacco = .31). Estimated power to detect a moderate treatment effect - 20% reduction in risk of initiation - exceeded 80% across all effect-size specifications tested.

Mixed model analyses (MM) will be used to examine effects on all outcomes, including primary outcomes (youth substance use and suicide, adult substance use) and secondary outcomes (proximal mediators of risk for primary outcomes). MM analyses will account for correlated observations within participants over time and examine intervention effects averaged across the entire post-program data collection period and at each post-program assessment point individually. Wave of data collection and Condition (TG or WW) X Wave interaction will be fixed effects. Time will be a repeated measures factor and study participant and family cluster will be included as random effects. After verifying that randomization yielded baseline equivalence across Conditions, the investigators will use either linear (ordinal/continuous outcomes) or generalized linear mixed models (dichotomous outcomes) to test Condition X Wave interactions. The overall difference between TG and WW groups across the follow-up period compared to baseline will be obtained by calculating the average of all 7 Condition X Wave interaction effects. These analyses will test hypotheses about immediate and sustained effects of intervention exposures on outcomes. Power estimates for MM analyses were calculated using GLIMMPSE software, specifying estimates of substance use at each wave derived from previous work with this population. Analyses indicate that the projected sample size will be sufficient to detect a small to moderate intervention effect - 20% reduction in substance use across time - with power greater than .80.

The final analytic approach will follow Muthén & Curran, estimating linear latent growth curve models (LGCM) to assess the effect of TG on outcome trajectories. The investigators will estimate the 'normative' trajectory of each outcome in the WW (comparison) group and the comparable trajectory in the TG (intervention) group. In the third step, the investigators will compare these trajectories and to determine whether there is a statistically significant change in the outcome trajectory related to TG intervention exposure. Finally, the investigators will evaluate the interaction between intervention exposure and initial level of the outcome to explore differential intervention effectiveness as a function of baseline levels for each outcome. Mplus Monte Carlo analyses were used to estimate power requirements for LGCM models and effect-size estimates were drawn from earlier etiological research. The power to detect slopes ranging from .14 to 1.4, were tested, estimating intercepts low (.05) consistent with our earlier findings and the young age of our study sample, setting alpha at .05, within each Condition group (TG treatment and WW comparison). Power estimates exceeded .90 to detect slope effects in all models.

ELIGIBILITY:
Inclusion Criteria:

* Youth participants:

  * 10-12 years old on the date of the first program session
  * Attending school on the reservation
  * Must enroll with an eligible adult
* Adult participants:

  * At least 18 years old
  * Must enroll with an eligible child
  * Must play a significant parenting role for the child enrolled in the study, as a parent, grandparent, other relative, legal guardian, or other household member.

Exclusion Criteria:

* Prisoners
* Decisionally-challenged adults

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Lifetime alcohol use | Change from baseline to 36 months after intervention
  Percentage reporting lifetime alcohol use (measured at baseline, post-test, and 6 month intervals for 36 months)
Alcohol initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported alcohol use
Past month frequency of any alcohol use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month alcohol use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month frequency of consumption of 4+ (for females) or 5+ (for males) alcoholic drinks at one time | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month alcohol consumption of 4+ drinks (for females) or 5+ (for males) (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month usual quantity of alcohol use [adults only] | Change from baseline to 36 months after intervention
  Trajectory of usual quantity of alcohol use in past month (# drinks, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime alcohol intoxication | Change from baseline to 36 months after intervention
  Percentage reporting lifetime alcohol intoxication (measured at baseline, post-test, and 6 month intervals for 36 months)
Alcohol intoxication initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported alcohol intoxication
Past month frequency of intoxication | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month alcohol intoxication (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime use of cough syrup (without parental permission) [youth only] | Change from baseline to 36 months after intervention
  Percentage reporting use of cough syrup (without parental permission) (measured at baseline, post-test, and 6 month intervals for 36 months)
Cough syrup use initiation (without parental permission) [youth only] | Up to 16 years of age
  Age of first reported non-medical cough syrup use
Past month frequency of use of cough syrup without parental permission [youth only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month use of cough syrup without parental permission (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month quantity of use of cough syrup without parental permission [youth only] | Change from baseline to 36 months after intervention
  Trajectory of quantity of past month cough syrup used without parental permission (1 or 2 teaspoons (0); ¼ of the bottle (1); ½ of the bottle (2); One whole bottle (3); More than one bottle (4); measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime marijuana use | Change from baseline to 36 months after intervention
  Percentage reporting lifetime marijuana use (measured at baseline, post-test, and 6 month intervals for 36 months)
Marijuana initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported marijuana use
Past month frequency of marijuana use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month marijuana use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime cigarette use | Change from baseline to 36 months after intervention
  Percentage reporting lifetime cigarette use (measured at baseline, post-test, and 6 month intervals for 36 months)
Cigarette initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported cigarette use
Past month frequency of cigarette use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month cigarette use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime use of electronic vapor products | Change from baseline to 36 months after intervention
  Percentage reporting use of electronic vapor products (measured at baseline, post-test, and 6 month intervals for 36 months)
Electronic vapor products initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported electronic vapor product use
Past month frequency of electronic vapor product use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month electronic vapor product use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime chewing tobacco use | Change from baseline to 36 months after intervention
  Percentage reporting chewing tobacco use (measured at baseline, post-test, and 6 month intervals for 36 months)
Chewing tobacco initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported chewing tobacco use
Past month frequency of chewing tobacco use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month chewing tobacco use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime inhalant use | Change from baseline to 36 months after intervention
  Percentage reporting inhalant use (measured at baseline, post-test, and 6 month intervals for 36 months)
Inhalant use initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported inhalant use
Past month frequency of inhalant use | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month inhalant use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime prescription pain medicine use without a prescription or other than as prescribed [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Percentage reporting non-medical use of prescription pain medicine (measured at baseline, post-test, and 6 month intervals for 36 months)
Prescription pain medicine use (non-medical) initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported non-medical prescription pain medicine use
Lifetime frequency of prescription pain medicine use without a prescription or other than as prescribed [adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of lifetime non-medical pain medicine use (# times, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month frequency of prescription pain medicine use without a prescription or other than as prescribed [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month non-medical prescription pain medicine use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime cocaine use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Percentage cocaine use (measured at baseline, post-test, and 6 month intervals for 36 months)
Cocaine use initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported cocaine use
Lifetime frequency of cocaine use [adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of lifetime cocaine use (# times, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month frequency of cocaine use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month cocaine use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime methamphetamine use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Percentage methamphetamine use (measured at baseline, post-test, and 6 month intervals for 36 months)
Methamphetamine use initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported methamphetamine use
Lifetime frequency of methamphetamine use [adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of lifetime methamphetamine use (# times, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month frequency of methamphetamine use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month methamphetamine use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime heroin use [adults only] | Change from baseline to 36 months after intervention
  Percentage heroin use (measured at baseline, post-test, and 6 month intervals for 36 months)
Heroin use initiation | Up to 16 years of age for youth; up to 30 years for adults
  Age of first reported heroin use
Lifetime frequency of heroin use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of lifetime heroin use (# times, measured at baseline, post-test, and 6 month intervals for 36 months)
Past month frequency of heroin use [youth aged 13+ and adults only] | Change from baseline to 36 months after intervention
  Trajectory of frequency of past month heroin use (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Lifetime suicidal ideation [youth only] | Change from baseline to 36 months after intervention
  Youth Risk Behavior Survey, middle school version, adapted to lifetime (ever seriously thought about suicide, ever made a plan, ever attempted); scored 0 to 3.
Past month suicidal ideation [youth only] | Change from baseline to 36 months after intervention
  Youth Risk Behavior Survey items adapted to past month time frame; Middle school version for youth up to age 12 (scored 0-3); High school version for youth aged 13+ (scored 0-8).

SECONDARY OUTCOMES:
Parent communication about alcohol and drugs [youth and adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of communication (measured at baseline, post-test, and 6 month intervals for 36 months)
Parent rules about substance use [youth and adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of setting rules about substance use (measured at baseline, post-test, and 6 month intervals for 36 months)
Substance use attitudes [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of attitudes (measured at baseline, post-test, and 6 month intervals for 36 months)
Substance use norms [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of norms (measured at baseline, post-test, and 6 month intervals for 36 months)
Antisocial behavior [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of behaviors (measured at baseline, post-test, and 6 month intervals for 36 months)
Association with deviant peers [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of association (measured at baseline, post-test, and 6 month intervals for 36 months)
Substance use resistance skills [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of skills (measured at baseline, post-test, and 6 month intervals for 36 months)
Substance use patterns (use of substances around children) [adults only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of patterns (measured at baseline, post-test, and 6 month intervals for 36 months)
Children's Hope Scale [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean scores, range 1-6, higher scores represent greater hope (measured at baseline, post-test, and 6 month intervals for 36 months)
Awareness of Connectedness scale (adapted) [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean scores, range 1-5, higher scores represent greater connectedness (measured at baseline, post-test, and 6 month intervals for 36 months)
Past week depression [youth only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean scores, range 1-4, higher scores represent greater depression (measured at baseline, post-test, and 6 month intervals for 36 months)
Family cohesion [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater cohesion (measured at baseline, post-test, and 6 month intervals for 36 months)
Family cohesion [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater cohesion (measured at baseline, post-test, and 6 month intervals for 36 months)
Family conflict [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater conflict (measured at baseline, post-test, and 6 month intervals for 36 months)
Family conflict [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater conflict (measured at baseline, post-test, and 6 month intervals for 36 months)
Family expressiveness [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater expressiveness (measured at baseline, post-test, and 6 month intervals for 36 months)
Family expressiveness [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean score, range 1-5, higher scores represent greater expressiveness (measured at baseline, post-test, and 6 month intervals for 36 months)
Use of family meetings [adult reports only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of use of family meetings (measured at baseline, post-test, and 6 month intervals for 36 months)
General parent-child communication [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of communication (measured at baseline, post-test, and 6 month intervals for 36 months)
General parent-child communication [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of communication (measured at baseline, post-test, and 6 month intervals for 36 months)
Parent warmth [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of warmth (measured at baseline, post-test, and 6 month intervals for 36 months)
Parent warmth [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of warmth (measured at baseline, post-test, and 6 month intervals for 36 months)
Parent negative affect [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of negative affect (measured at baseline, post-test, and 6 month intervals for 36 months)
Parent negative affect [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of negative affect (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental monitoring [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of monitoring (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental structure/rule setting [adult reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental structure/rule setting [youth reports] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental support of autonomy [youth report only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of support (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental use of discipline [adult report only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of discipline (measured at baseline, post-test, and 6 month intervals for 36 months)
Parental anger management [adult report only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of anger management (measured at baseline, post-test, and 6 month intervals for 36 months)
Support for parenting [adult report only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of support (measured at baseline, post-test, and 6 month intervals for 36 months)
Parenting self-efficacy [adult report only] | Change from baseline to 36 months after intervention
  Trajectory of change in mean reports of self-efficacy (measured at baseline, post-test, and 6 month intervals for 36 months)

OTHER OUTCOMES:
Daily fruit and vegetable consumption | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of daily consumption (# servings, measured at baseline, post-test, and 6 month intervals for 36 months)
Weekly physical activity | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of weekly physical activity (# days, measured at baseline, post-test, and 6 month intervals for 36 months)
Daily water consumption | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of daily water consumption (# glasses, measured at baseline, post-test, and 6 month intervals for 36 months)
Daily sugary drink consumption | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of daily water consumption (# drinks, measured at baseline, post-test, and 6 month intervals for 36 months)
Depression [adults only] | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of mean depression (measured at baseline, post-test, and 6 month intervals for 36 months)
Life satisfaction [adults only] | Baseline, post-test (1 week post-intervention), follow-up at 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Trajectory of change in reports of mean satisfaction (measured at baseline, post-test, and 6 month intervals for 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Whitesell, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
This study, conducted on an American Indian reservation, is under the oversight of the tribal Research Review Board (RRB). Representing a sovereign tribal nation, the RRB asserts ownership of data and limits how data can be used and shared. To ensure compliance with RRB requirements, the Data Access Committee (DAC) at the Centers for American Indian and Alaska Native Health at the University of Colorado Anschutz Medical Campus will manage data access. The DAC has a detailed process to ensure compliance with RRB protocol. Users will be required to sign data use agreements stipulating commitment to: 1) abide by all tribal research review requirements, including obtaining approval for secondary analysis before accessing data and following review procedures for dissemination; 2) use data only for approved research; 3) protect individual and, if relevant, community confidentiality; 4) secure data using appropriate computer technology; 5) destroy or return data after analyses are complete.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anticipated availability in late 2024, for a period of at least 5 years.
Access Criteria: See Plan Description for details of access requests through Data Access Committee.
URL: http://www.ucdenver.edu/academics/colleges/PublicHealth/research/centers/CAIANH/projects/Pages/DataAccessCommittee.aspx

REFERENCES:
- [Background] Ivanich JD, Mousseau AC, Walls M, Whitbeck L, Whitesell NR. Pathways of Adaptation: Two Case Studies with One Evidence-Based Substance Use Prevention Program Tailored for Indigenous Youth. Prev Sci. 2020 Jan;21(Suppl 1):43-53. doi: 10.1007/s11121-018-0914-5. PMID 29876790
- [Background] Whitesell NR, Mousseau AC, Keane EM, Asdigian NL, Tuitt N, Morse B, Zacher T, Dick R, Mitchell CM, Kaufman CE. Integrating Community-Engagement and a Multiphase Optimization Strategy Framework: Adapting Substance Use Prevention for American Indian Families. Prev Sci. 2019 Oct;20(7):1136-1146. doi: 10.1007/s11121-019-01036-y. PMID 31376058